CLINICAL TRIAL: NCT02894970
Title: A New Device for Measuring of Lung Photoplethysmography and Pulmonic Arterial Saturation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Israel Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: lung photoplethysmography
Record Dates: First submitted 2016-08-25; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Patent Ductus Arteriosus; Pulmonary Hypertension
MeSH Terms: conditions — Ductus Arteriosus, Patent; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Healthy adults: Healthy adults for checking feasibility of Pulmonary PPG
  Interventions: Device: Pulmonary PPG
- Healthy children: Healthy children for checking feasibility of Pulmonary PPG
  Interventions: Device: Pulmonary PPG
- Healthy neonates: Healthy neonates for checking feasibility of Pulmonary PPG and in order to be a control group for neonates with pulmonary hypertension.
  Interventions: Device: Pulmonary PPG
- Healthy preterm neonates: Healthy preterm neonates for checking feasibility of Pulmonary PPG and in order to be a control group for premature neonates with patent ductus arteriosus (PDA).
  Interventions: Device: Pulmonary PPG
- Preterm neonates with PDA: Preterm neonates with hemodynamic significant PDA. Intervention: evaluate Pulmonary PPG and oxygen saturation as compared to normal newborns.
  Interventions: Device: Pulmonary PPG
- Neonates with pulmonary hypertension: Neonates with pulmonary hypertension. Intervention: evaluate Pulmonary PPG and oxygen saturation as compared to normal newborns.
  Interventions: Device: Pulmonary PPG

INTERVENTIONS:
Device: Pulmonary PPG — Five minutes check with a lights source with two wave lengths of infrared and a detector.

SUMMARY:
To evaluate feasibility of photoplethysmography (PPG) of pulmonary arteries in adults children and neonates and to compare normal controls to premature newborns suffering from patent ductus arteriosus and neonates suffering from pulmonary hypertension.

DETAILED DESCRIPTION:
This study aims to check a new device for measuring lung photoplethysmography (PPG) of pulmonary arteries by delivering light through the chest wall. The aim is to evaluate pulmonary arteries' elasticity and oxygen saturation.

We will study adults children and neonates. We will study 20 healthy adults, 20 healthy children aged 2-8 years, twenty healthy neonates, 20 preterm neonates with patent ductus arteriosus (PDA) and 20 preterm neonates with no PDA. We will study also 20 neonates with pulmonary hypertension.

Each participant will be examined for 5 minutes and PPG signal will be recorded in a computer and evaluated offline later on. Pulmonic saturation will be calculated from absorption difference between two wave lengths of infrared light that will be used.

Our hypothesis is that the mentioned clinical conditions will affect PPG signal and pulmonary arterial oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamic stability

Exclusion Criteria:

* hemodynamic instability

Ages: 1 Day to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy volunteer adults and children, normal newborns, normal premature newborns and newborns suffering from patent ductus arteriosus and pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
difference in PPG or pulmonary saturation between conditions | 1 year

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nitzan M, Nitzan I. Pulse oximetry in the pulmonary tissue for the non-invasive measurement of mixed venous oxygen saturation. Med Hypotheses. 2013 Aug;81(2):293-6. doi: 10.1016/j.mehy.2013.04.026. Epub 2013 May 13. PMID 23679994